CLINICAL TRIAL: NCT00877734
Title: Phase IIIa Trial of Baclofen for Alcohol Dependence
Brief Title: Efficacy and Tolerability of Baclofen for Alcohol Dependence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: James C. Garbutt, MD/Principal Investigator, UNC Department of Psychiatry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: baclofen-unc-0507
Record Dates: First submitted 2008-02-07; First posted 2009-04-08 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2011-04

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; baclofen; pharmacotherapy; women
MeSH Terms: conditions — Alcoholism | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Baclofen
  Interventions: Drug: baclofen; Behavioral: BRENDA counseling
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo; Behavioral: BRENDA counseling

INTERVENTIONS:
Drug: baclofen — 10 mg Baclofen administered tid for 11 weeks
  Other Names: Lioresal
  Arms: 1
Drug: placebo — Placebo administered tid for 11 weeks
  Arms: 2
Behavioral: BRENDA counseling

SUMMARY:
This is a study of the efficacy and safety of baclofen for alcohol dependence. 80 outpatient subjects with DSM-IV alcohol dependence will be randomized to 10 mg three times a day (tid) baclofen or tid placebo. An effort will be made to recruit 40 men and 40 women. Subjects will receive BRENDA counseling over the 12 weeks of the trial. The Timeline Followback (TLFB) method will be used to assess drinking patterns. The primary outcome is % heavy drinking during the trial.

DETAILED DESCRIPTION:
The study will explore the efficacy and tolerability of a 12-week regimen of 10 mg t.i.d. baclofen vs. placebo in conjunction with behavioral therapy for reducing heavy drinking in 80 alcohol dependent individuals. Prior studies (Addolorato et al. 2000, 2002; Flannery et al., 2004) have found that baclofen reduces self-reported anxiety and craving; therefore, the proposed study also will assess baclofen's ability to reduce symptoms of these affective states. Furthermore, in our pilot study (Flannery et al, 2004), women appeared to respond more consistently than men, and therefore the study will also be balanced by gender.

ELIGIBILITY:
Inclusion Criteria

1. Men and women between the ages of 18 and 60 meeting DSM-IV criteria for current alcohol dependence.
2. Must have had at least 2 heavy drinking days (men > 5 drinks/days; women > 4 drinks/day) per week, on average and an average overall consumption of 21 drinks/week or more for men and 14 drinks/week or more for women during the 4 weeks prior to screening.
3. Able to understand and sign written informed consent.
4. Must be willing to refrain from drinking for three days prior to randomization day.
5. Express a desire to achieve abstinence or to greatly reduce alcohol consumption.
6. Must have a stable residence and be able to identify an individual who could locate subject if needed.

Exclusion Criteria

1. Clinically significant medical disease that might interfere with the evaluation of the study medication or present a safety concern (e.g., cirrhosis, kidney impairment, unstable hypertension, hypotension, diabetes mellitus, seizure disorder).
2. Clinically significant psychiatric illness including any psychotic disorder, bipolar disorder, or severe depression; suicidal ideation; substance use disorder other than alcohol or nicotine dependence or cannabis abuse.
3. History of complicated alcohol withdrawal, i.e. withdrawal seizure or delirium tremens.
4. Concurrent use of any psychotropic medication including antidepressants, mood stabilizers, antipsychotics, anxiolytics, stimulants, or hypnotics. However, subjects who have been on stable doses of the antidepressants fluoxetine, sertraline, paroxetine, citalopram, ecitalapram, trazodone or venlafaxine for two months will be eligible. Subjects who have been taking benzodiazepines for alcohol detoxification will be required to have a washout period of at least five half-lives (approximately 5 days) from those medications before being randomized.
5. Concurrent use of anticonvulsants, insulin, or oral hypoglycemics.
6. AST, or ALT > 3 times Upper Limit of Normal (ULN), or bilirubin > ULN, or creatinine > ULN.
7. Positive urine toxicology screen with the exception of cannabis. Individuals with positive cannabis screens will be excluded only if they have a history of cannabis dependence.
8. Pregnant women and women of childbearing potential who do not practice a medically acceptable form of birth control (oral or depot contraceptive, or barrier methods such as diaphragm or condom with spermicidal).
9. Women who are breastfeeding.
10. Individuals requiring inpatient treatment or more intense outpatient treatment for their alcohol dependence.
11. Participation in any clinical trial within the last 60 days.
12. Court-mandated participation in alcohol treatment or pending incarceration.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-04; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
% heavy drinking days | 2 years

SECONDARY OUTCOMES:
% relapse | 2 years
% abstinent days | 2 years
depression symptoms | 2 years
anxiety symptoms | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James C Garbutt, MD, Principal Investigator — UNC Department of Psychiatry
Locations (1):
- University of North Carolina at Chapel Hill School of Medicine, Chapel Hill, North Carolina, United States